CLINICAL TRIAL: NCT06141278
Title: China Hypertension and Diabetes Care Cascade Study
Acronym: CHICCs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Xuejun Yin, Dr., Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023026
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Hypertension; Diabetes
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Stakeholder-based participatory research will be conducted after CFIR-ERIC mapping activities to focus on partnerships, engagement, co-learning, and developing interventions incorporating interventions on existing practices. Three workshops will be held to reach agreements on the intervention tools, the implementation structure, the data collection procedures and the study audit process among the research team, local policymakers, and implementers. The participants and contents of each workshop are shown in Table 1. At the end of the workshop series, the implementation team from each county prepared a proposed intervention plan describing the steps needed to achieve their goals within a set timeline. The agreed plan of action considered their constraints and how to overcome those barriers.
  Interventions: Behavioral: Care cascade intervention
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Care cascade intervention — Co-designed integrated care based on the Chronic Care Model to improve hypertension and diabetes care cascade
  Arms: Intervention

SUMMARY:
This implementation study aims to identify priorities and formulate strategies to overcome health service delivery bottlenecks associated with hypertension and diabetes in rural China. Leveraging implementation frameworks, the study seeks to unravel the complexities embedded within the care cascade, paving the way for targeted interventions. Addressing the nuanced dynamics of the care cascade, this research will provide indispensable insights for optimising healthcare delivery in resource-limited settings, ultimately informing global perspectives on chronic disease management.

The overall aim of this study is to enhance the control of hypertension and diabetes in rural China through a systematic assessment and improvement of the care cascade, specifically:

1. To describe the cascade gap and identify barriers and facilitators at each cascade stage.
2. To develop practical interventions through stakeholder co-design.
3. To assess the effectiveness of developed interventions and evaluate implementation strategies.

DETAILED DESCRIPTION:
Hypertension and type 2 diabetes present substantial challenges to the Chinese health system. A nationwide survey revealed a hypertension prevalence of 37.2% among Chinese adults over 35, with only 44.7% aware of their diagnosis and a mere 30.1% receiving antihypertensive treatment, resulting in an overall control rate of 7.2% [1]. Similarly, diabetes prevalence in 2018 stood at 12.9%, with awareness and treatment rates of 37% and 33%, respectively [2]. Achieving hypertension and diabetes control is conditional on successful progression through screening, diagnosis, management, and control-a continuum demanding care continuity. The care cascade analysis, originally devised for communicable diseases (i.e., HIV and tuberculosis), offers a systematic approach that dissects disease management into a series of interconnected service delivery stages [3, 4]. This method evaluates patient progression, unveiling critical drop-offs between each stage. Despite existing population-based surveys detailing the awareness, prevalence and treatment of hypertension and diabetes in China, few studies provide a systematic diagnosis of what happens between stages and devise interventions tailored to each stage of the care cascade.

This implementation study aims to identify priorities and formulate strategies to overcome health service delivery bottlenecks associated with hypertension and diabetes in rural China. Leveraging implementation frameworks, the study seeks to unravel the complexities embedded within the care cascade, paving the way for targeted interventions. Addressing the nuanced dynamics of the care cascade, this research will provide indispensable insights for optimising healthcare delivery in resource-limited settings, ultimately informing global perspectives on chronic disease management.

The overall aim of this study is to enhance the control of hypertension and diabetes in rural China through a systematic assessment and improvement of the care cascade, specifically:

1. To describe the cascade gap and identify barriers and facilitators at each cascade stage.
2. To develop practical interventions through stakeholder co-design.
3. To assess the effectiveness of developed interventions and evaluate implementation strategies.

This is a hybrid design implementation study using mixed methods and integrates diverse implementation theories, models, and frameworks. The theoretical model synthesises the process model, determinant framework, and evaluation framework under the theory of implementation science (Figure 1). The Consolidated Framework for Implementation Research (CFIR) framework identifies multilevel factors influencing implementation. The chronic care model (CCM) is used to inform intervention development. The RE-AIM (reach, effectiveness, adoption, implementation, maintenance) framework is used to assess interventions across multiple dimensions. Normalisation Process Theory (NPT) is applied to measure elements critical for successful implementation and integration into routine work.

The study will be conducted in Gongyi, Wugang and Weifang counties of China. Study sites are selected by the study team on the basis of their willingness to participate and their proximity to the research team.

This study comprises three phases: 1) context analysis and need assessment, 2) intervention development; and 3) implementation and evaluation.

In phase one, we will conduct qualitative interviews with policymakers, physicians, primary care health providers and patients. This exploration distill the current state of hypertension and diabetes care in selected counties, identifying determinants within health delivery functions. The Consolidated Framework for Implementation Research (CFIR) framework will guide the assessment, allowing for a nuanced understanding of the intricacies influencing care cascades.

Phase two will employ stakeholder-based participatory research to craft targeted interventions. Systematic assessments of barriers identified in phase one will inform this process, facilitated by the CFIR-ERIC tool for mapping potential strategies. The resultant priority actions and interventions will be collaboratively co-designed with local service providers, health administrators, and decision-makers, ensuring a tailored and contextually relevant approach.

In phase three, a rigorously designed cluster-randomized controlled trial will be implemented to discern longitudinal changes in hypertension and diabetes care. Forty-eight villages will undergo randomisation into intervention and control groups, employing a 1:1 allocation ratio. Intervention villages will enact strategies developed in phase two, while control villages maintain usual care. The intervention period spans one year. To assess study outcomes at the population level, we will draw two independent random samples comprising 150 participants aged 35 to 74 from each village before and after the intervention. Outcomes measured include patient-level clinical outcomes (i.e., between-group differences in SBP, HbA1c), system-level service outcomes (i.e., successful progression through steps of cascade), and implementation outcomes (i.e., reach, adoption, feasibility, fidelity). Baseline surveys, conducted prior to randomization, aim to blind study staff from intervention allocation. The follow-up survey, performed one year after intervention initiation, will involve participants identified in the baseline survey, supplemented by the recruitment of an additional random sample. Qualitative interviews with stakeholders will be conducted to discern barriers and facilitators encountered during intervention implementation. Furthermore, an economic evaluation from the health services perspective is planned to provide a comprehensive understanding of the intervention's impact on healthcare resource utilisation and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Permanent residents of the surveyed village (residing for more than six months each year).
* Age between 35 and 74 years old.

Exclusion Criteria:

* Individuals with severe mental disorders or communication barriers.
* Individuals planning to move out of the village within the next year.
* Expected life expectancy of less than one year.
* Pregnant or lactating individuals.
* Individuals who are currently away (i.e. hospitalized, or residing elsewhere) so that cannot participate in the survey.

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14400 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of blood pressure control at baseline and at 12 month | Baseline and at 12 month
  The proportion of hypertension patients who have achieved BP control. We defined control as BP < 140/90 mmHg or lower in complex cases, such as diabetes
Change of blood glucose control at baseline and at 12 month | Baseline and at 12 month
  The proportion of diabetes patients who have achieved HbA1c < 6.5%
Change of SBP at baseline and at 12 month | Baseline and at 12 month
  Blood pressure is measured after the participant has rested for at least 15 minutes. Blood pressure is measured at least three times at 3 minutes intervals using the appropriate cuff size and a Digital Automatic Blood Pressure Monitor

SECONDARY OUTCOMES:
Screening rate at baseline and at 12 month | Baseline and at 12 month
  Percent of population with high blood pressure who have had previously had blood pressure measured according to standards. And percent of population with Diabetes who have ever had a blood glucose test.
Diagnosis rate at baseline and at 12 month | Baseline and at 12 month
  1. The proportion of people with hypertension in the catchment area of interest who are diagnosed at the facility level, where a diagnosis of hypertension follows at least three measurements of BP on two or more health visits with a systolic BP of 140 mmHg or higher or a diastolic BP of 90 mmHg or higher.
  2. The proportion of people with diabetes in the catchment area of interest who have a fasting plasma glucose of 7.0 mmol/l (126 mg/dl) or higher, or have a random plasma glucose of 11.1 mmol/l (200 mg/dl) or higher, or have an HbA1c measurement of 6.5% or higher
Treatment rate at baseline and at 12 month | Baseline and at 12 month
  1. The proportion of people who initiate treatment for hypertension, remain in care, and are followed-up by their service provider. A patient was considered being monitored by the care provider if there was evidence of BP being measured and recorded every month.
  2. The proportion of people who initiate treatment for diabetes, remain in care, and are followed-up by their service provider. A patient was considered being monitored by the care provider if there was evidence of blood glucose being measured and recorded every 3 months.

REFERENCES:
- [Derived] Yin X, Wang Z, Yang J, Li J, Han S, Feng W, Liu Q, Li N, Zhang L, Ke J, Wei X, Zhang J, Sarrafzadegan N, Shao R. Improvement of Care Cascade for Hypertension and Diabetes in Rural China: Protocol for an Implementation Study. J Clin Hypertens (Greenwich). 2024 Dec;26(12):1466-1478. doi: 10.1111/jch.14918. Epub 2024 Nov 4. PMID 39494843